CLINICAL TRIAL: NCT02880917
Title: Effects of Combined Treatment With tDCS and Cognitive Training on Attention and Working Memory in Patients With Fibromyalgia
Brief Title: Effects of Combined Treatment With tDCS and Cognitive Training in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 140369
Record Dates: First submitted 2016-08-08; First posted 2016-08-26 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Fibromyalgia
Keywords: Attention; Memory (short and long-term); Conflict monitoring tasks; Verbal fluency
MeSH Terms: conditions — Fibromyalgia | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive training + tDCs-Active (Active Comparator): tDCs active left dorsolateral prefrontal cortex (2mA,20 min) and Cognitive training (20min) at the same time.
  Interventions: Device: tDCS-Active; Other: Cognitive training
- Cognitive training+ tDCs-Sham (Sham Comparator): tDCs Sham dorsolateral prefrontal cortex ((2mA,20 min) and Cognitive training (20min) at the same time.
  Interventions: Device: tDCS-Sham; Other: Cognitive training

INTERVENTIONS:
Device: tDCS-Sham — Sham tDCS will involve an identical electrode montage, with stimulation ceasing after a 30-second ramp-up period to provide equivalent scalp sensation.
  Arms: Cognitive training+ tDCs-Sham
Device: tDCS-Active — tDCS was delivered using the anode electrode positioned over the left dorsolateral prefrontal cortex (DLPFE) and the cathode electrode at supra orbital right region. The electrodes were placed into a 25-35 cm2 square sponge immersed in saline solution for better current conductivity. Current density used was 2 mA and electrodes attached to the scalp were sustained by rubber band.
  Arms: Cognitive training + tDCs-Active
Other: Cognitive training — . The cognitive training consisted of an online application of a Dual N-Back task .The Training will last for 8 days.

SUMMARY:
Chronic pain represents an important health problem responsible for decreases in quality of life, and is associated with great negative impact in society and economy. In many cases, its treatment does not reach therapeutic success causing health professionals and patients dissatisfaction. Chronic pain is also associated with somatization, hopelessness and catastrophizing thinking. These information processing includes sensorial, emotional and cognitive-appraisal thinking, which manifests the working of neural networks at cortical and sub-cortical levels. Attention and memory are a central aspect in the processing of pain modulation. Like in addictions (e.g. smoking, alcohol), chronic pain may debut with displacement in the focus of attention and alterations in the sensorial processing in the incentive-motivation tests. Considering that other studies have indicated that experimental and clinical pain is capable of modulating cognitive activities such as attention,memory and expectation, in this study the investigators will test whether cognitive training, tDCS, or the combination of both interventions decrease cognitive deficits associated with Fibromyalgia

DETAILED DESCRIPTION:
Will be included women aged between 18 and 65 years, chronic pain fibromyalgia according to the criteria of the American College of Rheumatology, pain unresponsive to analgesics such as paracetamol, acetylsalicylic acid, ibuprofen, Carisoprodol, Zanaflex (Tizanidine) and Codeine and give informed consent to participate after initial evaluation. Primary outcome is to Evaluate whether the tDCS associated with cognitive retraining technique is able to modulate attentional bias in fibromyalgia patients. Secondary outcomes are: compare the effect of active tDCS and sham in: Assessed with the Visual Analog Scale for 8 days, Functional capacity, Conditional pain modulation (CPM), Maximal Heat Pain tolerance,Catastrophic thinking,Serum levels of Brain Derived Neurotrophic Factor (BDNF), Beck Depression Inventory, forward and backward digit span( WAIS),Pittsburgh sleep quality and State-Trait Anxiety Inventory (STAI) test.

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* literate
* right-handed
* 18 to 65 years of age
* who meet the criteria of the American College of Rheumatology (ACR) for fibromyalgia.

Exclusion Criteria:

* Pregnant women
* Contraindications to tDCS
* Metal implant in the brain
* History of alcohol or drug abuse in the last six months
* History of neurological disorders
* Unexplained fainting
* Self-reports of head injury or momentary loss of awareness
* Neurosurgery.
* Will also be excluded patients who have decompensated systemic diseases and / or chronic inflammatory diseases (ex .: lupus, rheumatoid arthritis).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Evaluate whether the tdcs associated with cognitive training technique or the combination of both interventions decrease memory deficits associated with Fibromyalgia. | 8 days
  I will use the rey auditory-verbal learning test(RAVLT) to evaluate the memory functions of patients with fibromyalgia, before and after treatment with TDCS and cognitive training.

SECONDARY OUTCOMES:
Pain | 8 days
  Assessed with the Visual Analog Scale for 8 days
Scale Functional capacity--(Using The Brazilian Portuguese version of the Profile of Chronic Pain.) | 2 days
  Measurement of functional capacity pre and pos application tDCS with scale functional capacity in chronic pain.
Test -Conditional pain modulation (CPM) | 2 days-pre and pos application tDCS
  The protocol for heat pain threshold is repeated while the contralateral hand is placed on iced water. The pain due to heat and cold reported on a Visual Analog Scale are recorded.

OTHER OUTCOMES:
Maximal Heat Pain Tolerance | 2 days
  Assessed using quantitative sensory testing. Briefly, the thermode placed in subjects forearm is heated until subject reports maximum tolerated pain. A maximal temperature of 52 Celsius has been previously programmed for the device to stop and cool down in order to avoid unintended injuries
Pain catastrophizing thoughts | 2 days
  Measurement of catastrophic thinking pre and pos application tDCS with catastrophizing.The level of catastrophic thinking will be assessed by the Pain Catastrophizing Scale on Treatment scale.
Serum levels of Brain Derived Neurotrophic Factor (BDNF) | 2 days
  Measurement of serum levels of BDNF pre and pos application tDCS
Beck Depression Inventory | 2 days
  Measurement of Beck Depression Inventory pre and pos application tDCS
Pittsburgh sleep quality | 2 days
  Measurement of Pittsburgh sleep quality pre and pos application tDCS
State-Trait Anxiety Inventory (STAI) test. | 2 days
  Measurement of State-Trait Anxiety Inventory (STAI) test pre and pos application tDCS
Electroencephalogram/ event-related potential P300 | 2 days
  Evaluate event-related potential (P300) pre and pos application tDCS
Paced Auditory Serial Addiction Test(PASAT) | 2 days
  I will use the Paced Auditory Serial Addiction Test to evaluate the memory functions of patients with fibromyalgia, before and after treatment with TDCS and cognitive training.
Controlled Oral Word Association Test | 2 days
  I will use the Controlled Oral Word Association Test to evaluate the verbal fluency of patients with fibromyalgia, before and after treatment with TDCS and cognitive training.
Forward and backward digit span | 2 days
  I will use the forward and backward digit span to evaluate the working memory of patients with fibromyalgia, before and after treatment with TDCS and cognitive training.
Auditory Consonant Trigrams | 2 days
  I will use the Auditory Consonant Trigrams to evaluate the working memory of patients with fibromyalgia, before and after treatment with TDCS and cognitive training.

CONTACTS AND LOCATIONS:
Overall Officials: Wolnei Caumo, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided